CLINICAL TRIAL: NCT00005473
Title: Cardiovascular Disease Trends 1980-91--A Gender Specific Perspective
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4956; R29HL055448 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Stroke

SUMMARY:
To test hypotheses related to gender differences in cardiovascular mortality trends between 1980 and 1991 in two southeastern New England communities which were part of the Pawtucket Heart Health Program.

DETAILED DESCRIPTION:
BACKGROUND:

The Pawtucket Heart Health Program was a community-based research and demonstration project in cardiovascular disease prevention in the town of Pawtucket, Rhode Island and in the non-intervention comparison town of New Bedford, Massachusetts. The study was initiated by the NHLBI in August, 1980. See also Study 1022.

DESIGN NARRATIVE:

There were four major areas of analysis: 1) gender differences in trends from 1980 to 1991 in total event rates, hospital discharge rates, in-hospital case-fatality and out of hospital deaths for coronary heart disease (CHD) and stroke; 2) gender specific analyses of methodological issues which may affect the interpretation of morbidity and mortality surveillance data; 3) gender differences in the presentation, diagnosis, and treatment of CHD and stroke which may influence morbidity and mortality trends; and 4) gender differences in the association between population trends in risk factors and morbidity and mortality trends.

The study was conducted using morbidity and mortality data collected by the Pawtucket Heart Health Program between 1980 and 1993, and risk factor data obtained through biennial cross-sectional household health surveys conducted in random samples of residents in the two study communities. Morbidity and mortality data were obtained according to standardized epidemiologic surveillance methods. Hospitalized cases of coronary heart disease and stroke were identified through hospital discharge records and were validated using a standardized diagnostic algorithm based on data abstracted from medical records. Out-of-hospital deaths identified through death certificate data were validated using an algorithm based upon medical history data and information concerning the circumstances of death obtained from informant interviews.

Gender specific trends in both age-adjusted and age specific morbidity and mortality were compared. Trends in rates estimated from events classified according to ICD-9 discharge and death certificate codes were contrasted with those estimated from cases validated by standardized diagnostic algorithms. Data regarding circumstances of death and in-hospital treatment were assessed in relation to potential influences on morbidity and mortality trends. Absolute changes over time and average annual percent change over time were evaluated using linear and log-linear regression regression techniques. Other analytic methods included logistic regression and analysis of variance. Expected annual event rates in men and women were estimated from risk factor data using equations based upon accelerated failure time Weibull models, and the impact of risk factors on mortality rates was assessed by comparing predicted with actual rates.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-07; Study Completion 2001-06 (Actual)

REFERENCES:
- [Background] Derby CA, Lapane KL, Feldman HA, Carleton RA. Trends in validated cases of fatal and nonfatal stroke, stroke classification, and risk factors in southeastern New England, 1980 to 1991 : data from the Pawtucket Heart Health Program. Stroke. 2000 Apr;31(4):875-81. doi: 10.1161/01.str.31.4.875. PMID 10753991
- [Background] Derby CA, Lapane KL, Feldman HA, Carleton RA. Sex-specific trends in validated coronary heart disease rates in southeastern New England, 1980-1991. Am J Epidemiol. 2000 Feb 15;151(4):417-29. doi: 10.1093/oxfordjournals.aje.a010222. PMID 10695601
- [Background] Derby CA, Lapane KL, Feldman HA, Carleton RA. Possible effect of DRGs on the classification of stroke: implications for epidemiological surveillance. Stroke. 2001 Jul;32(7):1487-91. doi: 10.1161/01.str.32.7.1487. PMID 11441190